CLINICAL TRIAL: NCT07218016
Title: Accelerometer Measured Early Recovery After Prolapse Surgery
Brief Title: The AccelERate Trial
Acronym: AccelERate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: RTI International (Other); University of California, San Diego (Other); University of Chicago (Other); Duke University (Other); Women and Infants Hospital of Rhode Island (Other); University of Pennsylvania (Other); Kaiser Permanente (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PFDN-34P01_1; UG1HD069013 (NIH); UG1HD054214 (NIH); UG1HD041267 (NIH); UG1HD054241 (NIH); UG1HD110057 (NIH); UG1HD069010 (NIH); U24HD069031 (NIH)
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Pelvic Organ Prolapse; Pelvic Organ Prolapse (POP); Pelvic Organ Prolapse Vaginal Surgery; Pelvic Organ Prolapse, Patient Education
Keywords: accelerometer; Pelvic Organ Prolapse (POP); Post-operative Recovery; recovery activities
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention)
- Postoperative Exercise regimen (Active Comparator)
  Interventions: Behavioral: Postoperative Exercise regimen

INTERVENTIONS:
Behavioral: Postoperative Exercise regimen — The intervention arm will be instructed to perform 30 minutes of medium intensity exercise (vigorous enough to cause shortness of breath, but light enough to be able to maintain a conversation) starting on postoperative day 3 and continuing at least 5 times weekly for 6 weeks. Participants in the intervention group will be allowed to select their preferred physical activity, and the activity will be performed without supervision. Participants in the control group will be given typical postoperative instructions with gradual resumption of activity.
  Arms: Postoperative Exercise regimen

SUMMARY:
The AccelERate study will evaluate the physical recovery of patients who have undergone Pelvic Organ Prolapse (POP) surgery. This will be evaluated via a self-reported recovery questionnaire completed daily. Participants will wear an accelerometer device on their non-dominant wrist and be given either routine or exercise-focused postoperative instructions. The primary outcome will be a comparison of the number of days needed to reach self-reported "mostly recovered" status between randomly assigned instruction groups.

DETAILED DESCRIPTION:
The AccelERate Trial is a single-masked RCT to determine if a prescribed early exercise regimen during the postoperative period in women undergoing minimally invasive surgery (MIS) for POP is associated with quicker recovery compared to standard recommendations for postoperative activities. AccelERate will go beyond existing research and be the first to implement and quantitatively evaluate with accelerometer data a postoperative exercise regimen and its effects on recovery and pelvic floor symptoms. We will quantify postoperative activity as well as recovery using self-report, performance-based testing, and objective medical assessment. In this way, we will rigorously investigate the regimen's effect on postoperative recovery and pelvic floor outcomes. Given prior findings that women who resume physical activity early in the postoperative period report fewer pelvic floor symptoms than women restricted from activity, we hypothesize that an intervention designed to encourage physical activity in the postoperative period may even further improve recovery without impacting short- or long-term functional and anatomic outcomes. Thus, AccelERate has the potential to transform care for women with POP who will no longer be required to alter their lifestyle and the activities for which they are having surgery.

The intervention arm will be instructed to perform 30 minutes of medium-intensity exercise (vigorous enough to cause shortness of breath, but light enough to be able to maintain a conversation) starting on postoperative day 3 and continuing at least 5 times weekly for 6 weeks (modeled after recent surgical postoperative physical activity studies). The amount of physical activity is in line with the Center for Disease Control and Prevention (CDC) guidelines and has been utilized in previous postoperative exercise studies. Participants in the intervention group will be allowed to select their preferred physical activity, and the activity will be performed without supervision.

Participants in the control group will be given liberalized postoperative instructions with gradual resumption of activity. The decision to allow women to liberally resume activity following surgery was informed by previous postoperative activity recommendation studies in women undergoing prolapse surgery.

All participants will undergo a baseline surgical evaluation including a POP-Q exam and PFDI-20 and PFIQ-7, complete AAS and record their physical activity for one week. Baseline physical activity data will include objective, quantitative measurement of movement using the accelerometer during waking hours for seven days (not necessarily consecutive days), and 30-second sit to stand test (STS).

Following surgery on postoperative day 3, participants will resume wearing an accelerometer continuously during waking hours. Those randomized to prescriptive exercise arm will be instructed to complete 30 minutes of medium intensity exercise as recommended by CDC and log their activity and percent recovery. If participants cannot complete the exercises, they will be asked to explain why (pain, nausea, catheter in place, logistical constraints, time constraints). Participants will be queried every day via the mobile research app as to the recovery they feel they have achieved. When a participant records "mostly" or "completely" recovered on 2-consecutive occasions (allowing for skipped days), she will stop receiving alerts. The primary outcome will be number of days since surgery at which the participant first reports being mostly recovered, provided she confirms that status on the next consecutive occasion (allowing for skipped days).

Postoperative study data will be collected remotely from participants via the app until 12-weeks. Accelerometer data will be downloaded from the devices 2-, 6-, and 12-week visits. At 12 weeks and 1 year, participants will undergo an in-office evaluation (including examination) assessing anatomic and functional outcomes with a surgeon masked to study assignment. They will also complete the AAS, PFDI-20, PFIQ-7, Decisional Regret Scale, NRS and PGI-I. At the baseline, 12-week, and 1-year visits, research staff will collect the self-administered activity questionnaires. At all study visits, research staff will record any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent
* Ambulatory women undergoing laparoscopic, robotic, or vaginal reconstructive or obliterative surgery for apical prolapse
* POP-Q >= Stage III
* Willing to participate in a postoperative exercise regimen
* Able to read and consent in English or Spanish
* Willing and able to wear an accelerometer prior to and after surgery (including agreeing to the terms of service), use an electronic data capture software, and record daily events
* Willing and able to install and use study-related smartphone app(s)
* Anticipated hospital discharge <= postoperative day 1

Exclusion Criteria:

* Inability or unwillingness to adhere to the exercise intervention
* Contraindication to medium-intensity exercise
* Comorbidities preventing physical activity
* Planned abdominal approach with laparotomy

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Recovery Status | From Day 3 post operation to 12 weeks post operation OR until participant achieves Mostly Recovered Status, whichever occurs first.
  A participant will be considered "mostly recovered" if they report feeling "mostly" or "completely" recovered on 2 consecutive daily self-report occasions, allowing for skipped days. The primary outcome will be number of days since surgery at which the participant first reports feeling mostly recovered, provided they confirm that status on the next consecutive occasion.

SECONDARY OUTCOMES:
Adherence to Exercise | From baseline to 12 weeks post operation.
  To measure adherence to a prescribed early exercise regimen using accelerometry for 12 weeks postoperatively and to determine if there is a difference in activity based on accelerometer data at 2, 6, and 12 weeks postoperatively between women in the prescribed exercise regimen group versus those in the standard postoperative activity instruction group.
Change From Baseline PFDI-20 Score | From baseline to 12 weeks post operation
  The Pelvic Floor Distress Inventory (PFDI-20) is a 20-question, validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of an Overall scale (range: 0-300) comprised of 3 sub-scales:
  1. Pelvic Organ Prolapse Distress Inventory (range: 0-100),
  2. Colorectal Anal Distress Inventory (range: 0-100) and,
  3. Urinary Distress Inventory (range: 0-100). The range of responses for all questions is 1-4 with (1) Not at all, (2) Somewhat, (3) Moderately, and (4), Quite a bit. Subscale scores are calculated by multiplying the mean value of all questions answered by 25 for the subscale. The range of score for each subscale is: 0-100 with 0 (least distress) to 100 (most distress). The PFDI-20 is calculated as the sum of the three subscales. Lower scores indicate better function / fewer symptoms for the PFDI-20 scale. Change from baseline = (Week[2,6,12] Score - Baseline Score).
Change From Baseline PFIQ-7 Score | From baseline to 12 weeks post operation
  The Pelvic Floor Impact Questionnaire short form (PFIQ-7) measuring the impact of bladder, bowel, and vaginal symptoms on a woman's daily activities, relationships and emotions is composed of an overall score (range 0-300), 3 subscales (7 questions each): the Urinary Impact Questionnaire (UIQ; range 0-100), the Pelvic Organ Prolapse Impact Questionnaire (POPIQ; range 0-100), and the Colorectal-Anal Impact Questionnaire (CRAIQ; range 0-100). The range of responses on all questions is 0-3 with (0) Not at all ... (3), Quite a bit. Subscale scores are calculated by multiplying the mean value of all answered questions for a scale by 100 divided by 3. The range of scores for each subscale is: 0-100 with 0 (least negative impact) to 100 (most negative impact). The PFI-7Q is the sum of the three subscales. Lower scores indicate better function / fewer symptoms for the PFIQ-7 score. Change from baseline = (Week[2,6,12] - Baseline Score).
PGI-I Score | From 12 weeks post operation to 1 year post operation
  The Patient Global Impression of Improvement (PGI-I) is a patient-reported measure of perceived condition improvement with treatment, as assessed on a scale of 1 (very much better) to 7 (very much worse).
Change From Baseline AAS Score | From baseline to 12 weeks post operation
  The Activity Assessment Scale (AAS) is a standardized measure of functional activity. The score ranges from 0 to 100 with higher scores indicating greater functional activity. Change from baseline = (Week[2,6,12] - Baseline Score).
Change From Baseline NRS Score | From baseline to 12 weeks post operation
  The Numeric Rating Scale (NRS) is a one-question validated patient-reported measure that quantifies the intensity of a specific symptom or experience on a numeric scale, from 0 (no pain) to 10 (worst pain imaginable). Higher scores are worse.
Change From Baseline SSCT Score | From baseline to 12 weeks post operation
  The 30-Second Sit to Stand Chair Test (SSCT) is a validated measure of lower body strength and endurance used to assess fall risk and functional ability in adults, especially older adults. The number of times a participant is able of going from sitting to standing is recorded and compared to normalized scores.
DRS Score | From 12 weeks post operation to 1 year post operation.
  The Decisional Regret Scale (DRS) is a standardized assessment of treatment satisfaction. It asks subjects to reflect on a particular decision and then rate each item on a Likert scale from 1 (strongly agree) to 5 (strongly disagree). Higher scores are worse.
Anatomic Recovery | From baseline to 12 weeks following operation
  Pelvic Organ Prolapse Quantification System (POP-Q) sites (Aa, Ba, C, D, Ap, Bp) are measured in centimeters relative to the hymenal plane. Measurements include genital hiatus (GH), perineal body (PB), and total vaginal length (TVL). This outcome represents the change in measurements. Evaluated as change from baseline. Change from baseline = (Week[12] - Baseline Score).

OTHER OUTCOMES:
Longitudinal Outcomes - Change From Baseline PFDI-20 Score | Baseline to 1 year post-operation
  The Pelvic Floor Distress Inventory (PFDI-20) is a 20-question, validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of an Overall scale (range: 0-300) comprised of 3 sub-scales: 1. Pelvic Organ Prolapse Distress Inventory (range: 0-100), 2. Colorectal Anal Distress Inventory (range: 0-100), and 3. Urinary Distress Inventory (range: 0-100). The range of responses for all questions is 1-4 with (1) Not at all, (2) Somewhat, (3) Moderately, and (4), Quite a bit. Subscale scores are calculated by multiplying the mean value of all questions answered by 25 for the subscale. The range of score for each subscale is: 0-100 with 0 (least distress) to 100 (most distress). The PFDI-20 is calculated as the sum of the three subscales. Lower scores indicate better function / fewer symptoms for the PFDI-20 scale. Change from baseline = (Year 1 Score - Baseline Score).
Longitudinal Outcomes - Change From Baseline PFIQ-7 Score | Baseline to 1 year post-operation
  The Pelvic Floor Impact Questionnaire short form (PFIQ-7) measuring the impact of bladder, bowel, and vaginal symptoms on a woman's daily activities, relationships and emotions is composed of an overall score (range 0-300), 3 subscales (7 questions each): the Urinary Impact Questionnaire (UIQ; range 0-100), the Pelvic Organ Prolapse Impact Questionnaire (POPIQ; range 0-100), and the Colorectal-Anal Impact Questionnaire (CRAIQ; range 0-100). The range of responses on all questions is 0-3 with (0) Not at all ... (3), Quite a bit. Subscale scores are calculated by multiplying the mean value of all answered questions for a scale by 100 divided by 3. The range of scores for each subscale is: 0-100 with 0 (least negative impact) to 100 (most negative impact). The PFIQ-7 is the sum of the three subscales. Lower scores indicate better function / fewer symptoms for the PFIQ-7 score. Change from baseline = (Year 1 - Baseline Score).
Longitudinal Outcomes - Change From Baseline AAS Score | Baseline to 1 year post-operation
  The Activity Assessment Scale (AAS) is a is a standardized a measure of functional activity. The score ranges from 0 to 100 with higher scores indicating greater functional activity.
Longitudinal Outcomes - Change From Baseline NRS Score | Baseline to 1 year post-operation
  The Numeric Rating Scale (NRS) is a one-question validated patient-reported measure that quantifies the intensity of a specific symptom or experience on a numeric scale, from 0 (no pain) to 10 (worst pain imaginable). Higher scores are worse.
Longitudinal Outcomes - Change From Baseline SSCT Score | Baseline to 1 year post-operation
  The 30 Second Sit to Stand Chair Test (SSCT) is a validated measure of lower body strength and endurance used to assess fall risk and functional ability in adults, especially older adults. The number of times a participant is able of going from sitting to standing is recorded and compared to normalized scores.
Longitudinal Outcomes - Anatomic Recovery | Baseline to 1 year post-operation
  Pelvic Organ Prolapse Quantification System (POP-Q) sites (Aa, Ba, C, D, Ap, Bp) are measured in centimeters relative to the hymenal plane. Measurements include genital hiatus (GH), perineal body (PB), and total vaginal length (TVL). This outcome represents the change in measurements.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Kaiser Permanente -- San Diego, San Diego, California
  - University of California - San Diego, San Diego, California
  - University of Chicago, Chicago, Illinois
  - Duke University, Duke Division of Urogynecology and Reconstructive Pelvic Surgery, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown/ Women and Infants Hospital of Rhode Island, Division of Urogynecology and Reconstructive Pelvic Surgery, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study data will be made available through DASH
Supporting Information: Study Protocol
Time Frame: Plan to submit full study dataset after the study is completed.
Access Criteria: Access is managed by DASH.
URL: http://dash.nichd.nih.gov/

REFERENCES:
- [Background] Onerup A, Andersson J, Angenete E, Bock D, Borjesson M, Ehrencrona C, Fagevik Olsen M, Larsson PA, de la Croix H, Wedin A, Haglind E. Effect of Short-term Homebased Pre- and Postoperative Exercise on Recovery After Colorectal Cancer Surgery (PHYSSURG-C): A Randomized Clinical Trial. Ann Surg. 2022 Mar 1;275(3):448-455. doi: 10.1097/SLA.0000000000004901. PMID 33843798
- [Background] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033
- [Background] Sung VW, Kauffman N, Raker CA, Myers DL, Clark MA. Validation of decision-making outcomes for female pelvic floor disorders. Am J Obstet Gynecol. 2008 May;198(5):575.e1-6. doi: 10.1016/j.ajog.2007.12.035. Epub 2008 Mar 7. PMID 18313632
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Cook KF, Dunn W, Griffith JW, Morrison MT, Tanquary J, Sabata D, Victorson D, Carey LM, Macdermid JC, Dudgeon BJ, Gershon RC. Pain assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S49-53. doi: 10.1212/WNL.0b013e3182872e80. PMID 23479545
- [Background] Barber MD, Kenton K, Janz NK, Hsu Y, Dyer KY, Greer WJ, White A, Meikle S, Ye W. Validation of the activities assessment scale in women undergoing pelvic reconstructive surgery. Female Pelvic Med Reconstr Surg. 2012 Jul-Aug;18(4):205-10. doi: 10.1097/SPV.0b013e31825e6422. PMID 22777368
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Nygaard IE, Clark E, Clark L, Egger MJ, Hitchcock R, Hsu Y, Norton P, Sanchez-Birkhead A, Shaw J, Sheng X, Varner M. Physical and cultural determinants of postpartum pelvic floor support and symptoms following vaginal delivery: a protocol for a mixed-methods prospective cohort study. BMJ Open. 2017 Jan 10;7(1):e014252. doi: 10.1136/bmjopen-2016-014252. PMID 28073797
- [Background] Liebermann M, Awad M, Dejong M, Rivard C, Sinacore J, Brubaker L. Ambulation of hospitalized gynecologic surgical patients: a randomized controlled trial. Obstet Gynecol. 2013 Mar;121(3):533-537. doi: 10.1097/AOG.0b013e318280d50a. PMID 23635615
- [Background] Daskivich TJ, Houman J, Lopez M, Luu M, Fleshner P, Zaghiyan K, Cunneen S, Burch M, Walsh C, Paiement G, Kremen T, Soukiasian H, Spitzer A, Jackson T, Kim HL, Li A, Spiegel B. Association of Wearable Activity Monitors With Assessment of Daily Ambulation and Length of Stay Among Patients Undergoing Major Surgery. JAMA Netw Open. 2019 Feb 1;2(2):e187673. doi: 10.1001/jamanetworkopen.2018.7673. PMID 30707226
- [Background] Engel O, Haikin Herzberger E, Yagur Y, Hershko Klement A, Fishman A, Constantini N, Biron Shental T. Walking to a better future? Postoperative ambulation after cesarean delivery and complications: A prospective study. Int J Gynaecol Obstet. 2022 May;157(2):391-396. doi: 10.1002/ijgo.13815. Epub 2021 Jul 17. PMID 34214190
- [Background] Ganer Herman H, Kleiner I, Tairy D, Gonen N, Ben Zvi M, Kovo M, Bar J, Weiner E. Effect of Digital Step Counter Feedback on Mobility After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2020 Jun;135(6):1345-1352. doi: 10.1097/AOG.0000000000003879. PMID 32459426
- [Background] Ganer Herman H, Ben Zvi M, Kleiner I, Tairy D, Kuper Sason L, Bar J, Kovo M. Mobility following cesarean delivery: an observational study utilizing pedometers. J Matern Fetal Neonatal Med. 2020 Mar;33(5):774-779. doi: 10.1080/14767058.2018.1500549. Epub 2018 Sep 10. PMID 30196735
- [Background] Nygaard IE, Shaw JM. Physical activity and the pelvic floor. Am J Obstet Gynecol. 2016 Feb;214(2):164-171. doi: 10.1016/j.ajog.2015.08.067. Epub 2015 Sep 6. PMID 26348380
- [Background] Heiman J, Onerup A, Wessman C, Haglind E, Olofsson Bagge R. Recovery after breast cancer surgery following recommended pre and postoperative physical activity: (PhysSURG-B) randomized clinical trial. Br J Surg. 2021 Jan 27;108(1):32-39. doi: 10.1093/bjs/znaa007. PMID 33640941
- [Background] Chen YP, Kuo YJ, Hung SW, Wen TW, Chien PC, Chiang MH, Maffulli N, Lin CY. Loss of skeletal muscle mass can be predicted by sarcopenia and reflects poor functional recovery at one year after surgery for geriatric hip fractures. Injury. 2021 Nov;52(11):3446-3452. doi: 10.1016/j.injury.2021.08.007. Epub 2021 Aug 10. PMID 34404509
- [Background] Kortebein P, Symons TB, Ferrando A, Paddon-Jones D, Ronsen O, Protas E, Conger S, Lombeida J, Wolfe R, Evans WJ. Functional impact of 10 days of bed rest in healthy older adults. J Gerontol A Biol Sci Med Sci. 2008 Oct;63(10):1076-81. doi: 10.1093/gerona/63.10.1076. PMID 18948558
- [Background] Neufer PD. The effect of detraining and reduced training on the physiological adaptations to aerobic exercise training. Sports Med. 1989 Nov;8(5):302-20. doi: 10.2165/00007256-198908050-00004. PMID 2692122
- [Background] Mirskaya M, Lindgren EC, Carlsson IM. Online reported women's experiences of symptomatic pelvic organ prolapse after vaginal birth. BMC Womens Health. 2019 Oct 29;19(1):129. doi: 10.1186/s12905-019-0830-2. PMID 31664987
- [Background] Mueller MG, Collins SA, Lewicky-Gaupp C, Tavathia M, Kenton K. Restricted Convalescence Following Urogynecologic Procedures: 1-Year Outcomes From a Randomized Controlled Study. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):e336-e341. doi: 10.1097/SPV.0000000000000922. PMID 32947549
- [Background] Bochenska K, Hall E, Griffith JW, Kenton K, Alverdy A, Lewicky-Gaupp C, Mueller M. The Promise of PROMIS in Pelvic Organ Prolapse. Female Pelvic Med Reconstr Surg. 2019 Nov-Dec;25(6):426-429. doi: 10.1097/SPV.0000000000000685. PMID 30570502
- [Background] Mueller MG, Lewicky-Gaupp C, Collins SA, Abernethy MG, Alverdy A, Kenton K. Activity Restriction Recommendations and Outcomes After Reconstructive Pelvic Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2017 Apr;129(4):608-614. doi: 10.1097/AOG.0000000000001924. PMID 28277355
- [Background] Weir LF, Nygaard IE, Wilken J, Brandt D, Janz KF. Postoperative activity restrictions: any evidence? Obstet Gynecol. 2006 Feb;107(2 Pt 1):305-9. doi: 10.1097/01.AOG.0000197069.57873.d6. PMID 16449116
- [Background] Winkelman WD, Erlinger AL, Haviland MJ, Hacker MR, Rosenblatt PL. Survey of Postoperative Activity Guidelines After Minimally Invasive Gynecologic and Pelvic Reconstructive Surgery. Female Pelvic Med Reconstr Surg. 2020 Dec 1;26(12):731-736. doi: 10.1097/SPV.0000000000000697. PMID 30707119
- [Background] Anger JT, Mueller ER, Tarnay C, Smith B, Stroupe K, Rosenman A, Brubaker L, Bresee C, Kenton K. Robotic compared with laparoscopic sacrocolpopexy: a randomized controlled trial. Obstet Gynecol. 2014 Jan;123(1):5-12. doi: 10.1097/AOG.0000000000000006. PMID 24463657
- [Background] Romanova AL, Carter-Brooks C, Ruppert KM, Zyczynski HM. 30-Day unanticipated healthcare encounters after prolapse surgery: impact of same day discharge. Am J Obstet Gynecol. 2020 May;222(5):482.e1-482.e8. doi: 10.1016/j.ajog.2019.11.1249. Epub 2019 Nov 13. PMID 31733206
- [Background] Buckwalter JA. Activity vs. rest in the treatment of bone, soft tissue and joint injuries. Iowa Orthop J. 1995;15:29-42. PMID 7634042
- [Background] Carter-Brooks CM, Du AL, Ruppert KM, Romanova AL, Zyczynski HM. Implementation of a urogynecology-specific enhanced recovery after surgery (ERAS) pathway. Am J Obstet Gynecol. 2018 Nov;219(5):495.e1-495.e10. doi: 10.1016/j.ajog.2018.06.009. Epub 2018 Jun 18. PMID 29913175
- [Background] Nager CW, Visco AG, Richter HE, Rardin CR, Rogers RG, Harvie HS, Zyczynski HM, Paraiso MFR, Mazloomdoost D, Grey S, Sridhar A, Wallace D; NICHD Pelvic Floor Disorders Network. Effect of Vaginal Mesh Hysteropexy vs Vaginal Hysterectomy With Uterosacral Ligament Suspension on Treatment Failure in Women With Uterovaginal Prolapse: A Randomized Clinical Trial. JAMA. 2019 Sep 17;322(11):1054-1065. doi: 10.1001/jama.2019.12812. PMID 31529008
- [Background] Barber MD, Brubaker L, Burgio KL, Richter HE, Nygaard I, Weidner AC, Menefee SA, Lukacz ES, Norton P, Schaffer J, Nguyen JN, Borello-France D, Goode PS, Jakus-Waldman S, Spino C, Warren LK, Gantz MG, Meikle SF; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network. Comparison of 2 transvaginal surgical approaches and perioperative behavioral therapy for apical vaginal prolapse: the OPTIMAL randomized trial. JAMA. 2014 Mar 12;311(10):1023-34. doi: 10.1001/jama.2014.1719. PMID 24618964
- See also: Physical Activity Guidelines for Americans — https://health.gov/sites/default/files/2019-09/Physical_Activity_Guidelines_2nd_edition.pdf#page=56